CLINICAL TRIAL: NCT04701281
Title: Phase Ib/II Study of Intra-Arterial Liver Isolation Chemotherapy in Patients With Hepatic Metastases From Colorectal Cancer
Brief Title: Study of Intra-Arterial Oxaliplatin Plus Capecitabine to Treat Liver Metastases From Colorectal Cancer
Acronym: SYS-CAPLIOX
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding depleted to continue study
Sponsor: AllVascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS-CAPLIOX
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: liver; metastases; colon; rectal; intra-arterial
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Single arm, two cohorts:
  Cohort 1: 1st line patients, RAS mutant; Cohort 2: pre-treated or refractory patients, no specific mutation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-arterial LIOX + Capecitabine (Experimental): 5 - 7 LIOX (liver isolation oxaliplatin) intra-arterial infusions over 8 weeks + capecitabine
  Interventions: Combination Product: Intra-arterial LIOX + Capecitabine

INTERVENTIONS:
Combination Product: Intra-arterial LIOX + Capecitabine — 5 - 7 LIOX (liver isolation oxaliplatin) intra-arterial infusions over 8 weeks + capecitabine

SUMMARY:
The treatment proposed in this trial is to administer intra-arterial chemotherapy to liver metastases from colorectal cancer when the blood flow to and from the liver has been isolated via balloon catheters through a vascular access system called the AVAS. The objective of this study is to evaluate the tumour response of repeated and isolated intra-arterial liver isolation oxaliplatin compared with the standard systemic chemotherapy (intravenous 5-FU + leucovorin + oxaliplatin [FOLFOX] or oral capecitabine with IV oxaliplatin [XELOX]).

DETAILED DESCRIPTION:
The treatment proposed in this study is based on the hypothesis that direct arterial infusion of chemotherapy to metastatic tumours of the liver whilst the blood flow to the organ is isolated could potentially yield benefits that cannot be achieved with existing treatment regimens.

There are three treatment stages; implantation of a vascular access device (known as the AVAS), intra-arterial liver isolation oxaliplatin (LIOX) infusions and explantation of the AVAS.

Implantation: the participant is admitted to hospital and the AVAS is surgically implanted under general anaesthetic. The AVAS is an implantable large bore cannula with one end that can be anastomosed directly onto a peripheral vessel and the opposite end exiting the patient's skin. The device can be opened to access the patient's vasculature when required and closed when the device is not in use. In accordance with the manufacturer's Instructions-For-Use (IFU), the AVAS will be implanted in the axillary artery (i.e. the upper pectoral area) or in the common femoral artery (upper thigh) by a surgeon experienced in vascular disease. The implantation procedure takes around 2 hours. After implantation, the participant is monitored overnight.

Intra-arterial LIOX infusions: the participant is admitted to the angiography suite and under general anaesthetic or conscious sedation, intra-arterial hepatic isolation chemotherapy infusion is administered by an interventional radiologist. The first infusion can be administered 2 days after device implantation and infusions are spread out over an 8-week period at a maximum such that the patient receives 5 to 7 infusions in total, has at least 2 full calendar days between each infusion, and there are no more than 2 infusions over any 7 consecutive days. Each infusion can take between 2-3 hours during the first few infusions but should only take 1-2 hours for the remaining infusions as the radiologist becomes familiarised with the patient's vascular anatomy.

During the Phase Ib stage, the starting dose of the oxaliplatin infused will be 50mg/m^2 and this dose will be escalated by 10mg/m^2 with each patient until an optimal dose is established. The optimal dose will be used for all patients enrolled during the Phase II stage.

Explantation: the final infusion session is followed by the device explantation immediately, or at a later time depending on the availability of operating rooms and the condition of the participant. The surgical removal of the device takes approximately 1-2 hours, the participant is monitored overnight and discharged the next day.

In addition, capecitabine will be administered orally as per standard care (1000 mg/m^2 twice daily in 2 week cycles) throughout the study treatment period (from enrolment to 4 weeks after the AVAS explantation) as a form of systemic disease management. The oncologist may modify the capecitabine dose/frequency based on the patient's response to the medication.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 years or older, with hepatic metastases from histologically proven adenocarcinoma of the colon/rectum;
2. Limited extrahepatic metastases in the lung or lymph nodes;
3. Confirmed non-progressive disease in the liver, per RECIST v1.1, halfway into the first-line systemic chemotherapy regimen after a minimum of 4 cycles of FOLFOX/XELOX ± monoclonal antibodies OR liver-dominant pre-treated or refractory patients;
4. Genotype: RAS mutant for first line patients only. All genetic mutations allowable for pre-treated or refractory patients;
5. Prior treatment with monoclonal antibody treatment is ≥ 4 weeks before implantation;
6. Considered medically fit for repeated general anaesthesia;
7. ECOG performance status 0-1;
8. Adequate bone marrow function (within 14 days of enrolment):

   Haemoglobin ≥ 100 g/L; ANC ≥ 1.5 × 10^9/L; Platelet Count ≥ 100 × 10^9/L;
9. Adequate renal function (within 14 days of enrolment):

   Serum Creatinine ≤ 1.5 × Upper Limit of Normal;
10. Adequate liver function (within 14 days of enrolment):

    Bilirubin ≤2.0 × Upper Limit of Normal; AST ≤ 5 × Upper Limit of Normal;
11. Normal coagulation (within 14 days of enrolment):

    INR ≤ 1.5;
12. Able to understand the risks and benefits of the study and provide signed, written informed consent to participate;
13. Willing and able to comply with all study requirements and assessments;

Exclusion Criteria:

1. CT-angiogram confirms unsuitable vascular anatomy;
2. No measurable liver disease per RECIST v1.1;
3. Evidence of ascites, cirrhosis, portal hypertension, main portal venous tumour involvement or main portal venous thrombosis;
4. Allergies to contrast agents;
5. Previous hypersensitivity or laryngo-pharyngeal dysaesthesia associated with oxaliplatin;
6. Previous allergies associated with 5-FU or oxaliplatin;
7. Grade > 2 peripheral neuropathy (CTCAE 5.0);
8. Significant co-morbidities;
9. Life expectancy ≤ 3 months;
10. Pregnant or breastfeeding women, or women of childbearing potential and men who are not on a reliable form of birth control or barrier method of contraception;
11. Enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during this clinical study;
12. Medical conditions that preclude the testing required by the protocol, or limit study participation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Liver-specific response rate (RR) | 4 weeks post explantation of AVAS;
  Assessed via clinical imaging and tumour markers using RECIST v1.1;

SECONDARY OUTCOMES:
Two-year survival rate; | 3, 6, 9, 12, 18 and 24 months post end of treatment and AVAS explantation;
  During follow-up;
Progression free survival (PFS); | 3, 6, 9, 12, 18 and 24 months post end of treatment and AVAS explantation;
  During follow-up;
Systemic side effects to chemotherapy | From enrolment until primary outcome is assessed (4 weeks post AVAS explantation);
  Assessed by collection of adverse events using Common Terminology Criteria for Adverse Events (CTCAE v5.0);
Organ isolation capability | Measured after each infusion treatment, through study completion, up to 8 weeks;
  Determined by pressure readings on catheters;
Conversion to resection rate; | Assessed at end of treatment, 4 weeks post AVAS explanation;
Health-related Quality of life (QoL); | Through study completion, an average of 8 weeks;
  Assessed quality of life questionnaire : comprising of 28 lifestyle and health questions using a four point scale (not at all, a little, quite a bit, very much) and 2 questions measuring overall health and overall quality of life on a visual analogue scale (1 very poor - 7 excellent);
Health-related Quality of life (QoL); | Through study completion, an average of 8 weeks;
  Assessed via quality of life questionnaire : comprising 10 digestion and and health questions using a four point scale (not at all, a little, quite a bit, very much);

CONTACTS AND LOCATIONS:
Overall Officials: Nick Pavlakis, A/Prof, Study Chair — GenesisCare, St Leonards
Locations (5):
- Australia (5):
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - GenesisCare, St Leonards, Saint Leonards, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Sydney Southwest Private Hospital, Sydney, New South Wales
  - Gold Coast Private Hospital, Southport, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.allvascular.com/